CLINICAL TRIAL: NCT02494856
Title: Comparison of the Clinical Efficacy of Naproxen, Associated or Not With Esomeprazol, in the Control of Pain, Swelling and Trismus in Lower Third Molar Removal
Brief Title: Comparison of the Clinical Efficacy of Naproxen, Associated or Not With Esomeprazol, in Lower Third Molar Removal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Giovana Maria Weckwerth (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor-Investigator, Giovana Maria Weckwerth, DDS, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: CAAE: 30317314.4.0000.5417
Record Dates: First submitted 2015-07-07; First posted 2015-07-10 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Pain; Other Surgical Procedures; Impacted Third Molar Tooth
Keywords: Naproxen; Lower third molar; Oral Surgery; Esomeprazole
MeSH Terms: conditions — Pain | interventions — Surgical Procedures, Operative; Naproxen; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery with Naproxen (Experimental): Fifty healthy volunteers underwent removal of symmetrically positioned lower third molars, will be treated to control pain, swelling and trismus with naproxen 500mg.
  Interventions: Drug: Surgery with Naproxen
- Surgery with Naproxen and Esomeprazole (Experimental): Fifty healthy volunteers underwent removal of symmetrically positioned lower third molars, will be treated to control pain, swelling and trismus with naproxen 500mg and esomeprazole 20mg.
  Interventions: Drug: Surgery with Naproxen and Esomeprazole

INTERVENTIONS:
Drug: Surgery with Naproxen — After lower third molars surgeries, clinical efficacy of the Naproxen 500mg was study.
  Other Names: Lower third molar surgery with Naproxen
  Arms: Surgery with Naproxen
Drug: Surgery with Naproxen and Esomeprazole — After lower third molars surgeries, clinical efficacy of the Naproxen 500mg and Esomeprazole 20mg was study.
  Other Names: Lower third molar surgery with Naproxen and Esomeprazole
  Arms: Surgery with Naproxen and Esomeprazole

SUMMARY:
The present clinical trial randomized compared the clinical efficacy of the naproxen associated or not with esomeprazol, for the removal of lower third molars. Onset, duration of postoperative analgesia, duration of anesthetic action on soft tissues, intraoperative bleeding, hemodynamic parameters, postoperative mouth opening and wound healing at the 7th postoperative day were evaluated. For this purpose, 50 healthy volunteers underwent removal of symmetrically positioned lower third molars, in two separate appointments (one to two months apart), under local anesthesia with either articaine 4% (1:200,000 adrenaline) in a doubleblind, randomized and crossed manner.

DETAILED DESCRIPTION:
The control of pain, swelling and trismus in patients undergoing oral and maxillofacial surgery is frequently performed through the administration of non-steroidal antiinflammatory drugs (NSAIDS). Studies have shown that NSAIDS exert their therapeutic effect by the inhibition of cyclooxigenases (COX) 1 and 2, which determines the inhibition of prostaglandins production whose effects potentiate the action of many inflammatory mediators. The present study aims to evaluate in a double blind, randomized and cross over manner the clinical efficacy of naproxen (500 mg) and naproxen in association with esomeprazol (500 mg and 20 mg), both administered by oral route every 12 h during 4 days, in 50 patients aged 18 years or older that require removal of both lower third molars symmetrically positioned. The following parameters will be analyzed: 1) subjective postoperative pain evaluation, with the aid of a visual analogue scale, 2) mouth opening before the surgery, on the 2nd and 7th postoperative days (moment of suture removal), 3) beginning and duration of the surgery after anesthetic administration, 4) incidence, type and severity of adverse reactions, 5) total amount of rescue analgesic medication (paracetamol), 6) facial swelling measured on the 2nd and 7th postoperative days (in comparison with the measurements before the surgery). The comparative analyses of the data along with the application of the adequate statistical tests will provide the basis for an evaluation of the clinical efficacy of both NSAIDS.

ELIGIBILITY:
Inclusion Criteria:

* Need of lower third molar surgeries in similar positions

Exclusion Criteria:

* Presence of systemic diseases;
* Presence of local inflammation and/or infection;
* Any history of allergic reaction to local anesthetics, gastrointestinal bleeding or ulceration;
* Cardiovascular, kidney or hepatic diseases;
* Patients who are making use of antidepressants, diuretics or anticoagulants;
* Asthma and allergy to aspirin, naproxen or any other nonsteroidal antiinflammatory drug;
* Regular use of any nonsteroidal antiinflammatory drug,
* pregnancy or
* breast feeding.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of postsurgical pain | Seventh postoperative day
  Subjective evaluation of postsurgical pain, which was annotated by the volunteer, a Visual Analogue Scale (VAS, 0-100 mm) and total amount (mg) of rescue medication consumption in the postoperative period. The subjective pain evaluations will be performed by patients at the following times after administration of the drugs [0, 15, 30 and 45 min, 1; 1.5; 2; 3; 4; 5; 6; 7; 8; 10; 12; 16; 24 hr, 48, 72 and 96 h].
Quality of anesthesia | During the surgical procedure
  Quality of anesthesia during surgery based on a category 3point scale: 1) the patient reported no discomfort; 2) the patient reported discomfort, without the need to supplement the anesthesia; 3) reported some discomfort by the patient, requiring anesthesia complementation. Intraoral bleeding that will be evaluated by the surgeon according to a 3point scale (1: minimal, 2: normal and 3: Maximum), immediately after the following steps: injection of the first cartridge anesthesia, incision, mucoperiosteal detachment, osteotomies, tooth section, extraction, cleaning and suturing.
Intraoperative bleeding | During the surgical procedure
  Intraoperative bleeding, rated by the surgeon according to a 3 point category rating scale (1 minimal bleeding; 2 normal bleeding; 3 excessive bleeding) (SISK, 1986), immediately after the following steps: injection of the first cartridge of articaine, tissue incision, flap reflection, bone removal (when this procedure was necessary), tooth extraction, cleaning of the operated site, and completion of suturing.
Blood pressure | During the surgical procedure
  Systolic blood pressure, diastolic, and mean to be verified and recorded at surgical moments previously described (injection of the first cartridge anesthesia, incision, mucoperiosteal detachment, osteotomies, tooth section, extraction, cleaning and suturing), carried out with the aid of a system for monitoring hemodynamic parameters.
Heart rate | During the surgical procedure
  Heart rate to be verified and recorded surgical at moments described above, carried out with the aid of a system for monitoring hemodynamic parameters.
Oxygen saturation | During the surgical procedure
  Oxygen saturation to be verified and recorded at surgical moments described above, carried out with the aid of a system for monitoring hemodynamic parameters.

SECONDARY OUTCOMES:
Postoperative mouth opening | Second and Seventh postoperative days
  Mouth opening (mm) between the mesial-incisal corners of the upper and lower right central incisors at maximum opening of the jaws was measured and recorded before the surgery and during the second and seventh postoperative days.
Onset and duration of surgery after administration of anesthetic | During the surgery
  Will only be considered those surgeries in which there is no long time gap between the two surgical times.
Incidence, type and severity of adverse reactions | Seventh postoperative day
  Will be considered as adverse reactions: gastrointestinal irritation, nausea, vomiting, bleeding, allergy, headache, dizziness, drowsiness or any other type of reaction presented after surgery.
Total amount of rescue medication | Seventh postoperative day
  The total amount of rescue medication that was used by the patient during the postoperative period (paracetamol 750 mg) will be analyzed.
Measurement the facial edema | On the second day after surgery and on the seventh day after surgery.
  It will apply the method used by Ustun et al. (2003), which takes into account the sum of the following measures (obtained with flexible tape measure): A) distance between the lateral corner of the eye and the gonion, B) away from the tragus corner of the mouth and C) away from the tragus to the soft tissue of pogonion. Preoperative sum of three measures will be considered as the baseline that way. The difference between the values obtained in the postoperative period and baseline indicate the facial edema in the 2nd and 7th days.

CONTACTS AND LOCATIONS:
Overall Officials: Giovana M Weckwerth, DDS, Principal Investigator — 416.016.638-54
Locations (1):
- University of São Paulo, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No